CLINICAL TRIAL: NCT02389608
Title: The Immediate Effect of Electrical Stimulation Transcranial Direct Current (tDCS) Associated With the Use of FES, in Muscle Activity of the Tibialis Anterior Muscle, Balance and Plantar Pressure Distribution of Individuals With Hemiparesis Due to Stroke - Randomized, Double Blind
Brief Title: The Immediate Effect of Electrical Stimulation Transcranial Direct Current (tDCS) Associated With the Use of FES, in Muscle Activity of the Tibialis Anterior Muscle, Balance and Plantar Pressure Distribution of Individuals With Hemiparesis Due to Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Aline Marina Alves Fruhauf, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/18128-6
Record Dates: First submitted 2015-02-18; First posted 2015-03-17 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2015-11

CONDITIONS: STROKE
Keywords: Transcranial direct current stimulation; functional electrical stimulation; hemiparesis; electromyography; balance
MeSH Terms: conditions — Stroke; Paresis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1- tDCS 2--FES (Experimental): 1. Transcranial stimulation ( tDCS ) will be administered using Tct Research 1 CH tdcs Simulator model 101. tDCS will be performed for 20 minutes and intensity 2mA associated active contraction of the TA muscle. Placebo tDCS will follow the same procedures as active tDCS with active, but the tDCS device will only be switched on for 20 seconds.
  2. Functional electrical stimulation (FES) will be administered using QUARK® FES VIF 995 DUAL device. The duration of active FES will be 20 minutes, associated with active contraction of the TA muscle. The pulse width will be 250 µs, modulated at a frequency of 50 Hz, with one to two stimulation cycles (6 seconds on and 12 seconds off) and the intensity will be increased until reaching the motor threshold. Placebo FES will follow the same procedures as active FES , but the FES device will only be switched on for 20 seconds, following which the intensity will be gradually reduced to 0 mA.
  Interventions: Device: Transcranial direct current stimulation (tDCS); Device: Functional electrical stimulation (FES); Device: Sham stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — The active tDCS and placebo will be applied to the primary motor cortex (M1) and FES active and placebo will be applied to the anterior tibial muscle (TA).
Device: Functional electrical stimulation (FES)
Device: Sham stimulation

SUMMARY:
Background: Transcranial direct current stimulation (tDCS) is currently considered a beneficial method for patients with neurological problems due to the modulation of cortex activity as well as the enhancement and prolongation of functional gains achieved during physical therapy. Purpose: The aim of the proposed study is to evaluate the immediate effects of a session of tDCS over the primary motor cortex combined with functional electrical simulation (FES) on electrical activity of the tibialis anterior muscle, balance and distribution of plantar pressure in individuals with hemiparesis stemming from a stroke. A further aim is to determine whether the effects of the combination of both stimulation methods are better than those achieved when each method is employed alone. Methods/design: A randomized, double-blind, crossover, cross-sectional study will be conducted involving 30 stroke survivors with hemiparesis who meet the eligibility criteria. Evaluations will involve an identification and screening chart, the classification of motor impairment using the Fugl-Meyer Scale, the determination of spasticity of the triceps surae muscle (modified Ashworth scale), electromyography of the tibialis anterior muscle, static balance and cognitive dual-task balance (stabilometry) and plantar pressure. After the initial evaluations, the participants will undergo four interventions: 1) anodal tDCS + placebo FES + active tibialis anterior contraction; 2) placebo tDCS + active FES + active tibialis anterior contraction; 3) anodal tDCS + active FES + active tibialis anterior contraction; and 4) placebo tDCS + placebo FES placebo + active tibialis anterior contraction. tDCS will be administered over the primary motor cortex and FES will be administered over the tibialis anterior muscle. The order of the different protocols will be randomized and both the evaluator and patients will be blinded to which protocol is being administered.

ELIGIBILITY:
Inclusion criteria:

* 30 individuals with hemiparesis stemming from a stroke;
* Either gender;
* Able to maintain a standing position without an assistance device for at least 60 seconds;
* Signed statement of written consent.

Exclusion criteria:

* Adverse health condition (beyond hemiparesis) that affects balance;
* Use of medication that can affect balance;
* Positive cutoff point for cognitive deficit (Mini Mental State Examination);
* Illiteracy;
* Wernicke's aphasia;
* Reduced ankle mobility due to history of ankle fracture and use of pins in ankle;
* TA muscle strength less than grade 1;
* Contraindication for tDCS (history of recurrent seizures, recurrent epilepsy and brain tumor in stimulation site);
* Skin infection at tDCS and/or FES site;
* Anesthesia or hyperesthesia at FES site.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
electromyography (EMG ) activity of Tibialis Anterior Muscle. | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411